CLINICAL TRIAL: NCT00021554
Title: A Phase III Open-Label, Randomized, Active-Controlled Study Assessing the Efficacy and Safety of T-20 (HIV-1 Fusion Inhibitor) in Combination With an Optimized Background Regimen, Versus Optimized Background Regimen Alone, in Patients With Prior Experience and/or Prior Documented Resistance to Each of the Three Classes of Approved Antiretrovirals (Nucleoside Reverse Transcriptase, Non-Nucleoside Reverse Transcriptase and Protease Inhibitors)
Brief Title: T-20 in HIV Patients With Prior Drug Treatment and/or Resistance to Each of the Three Classes of Anti-HIV Drugs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Trimeris (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 295D; T20-302
Record Dates: First submitted 2001-07-21; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-05

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; HIV Protease Inhibitors; RNA, Viral; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; pentafuside
MeSH Terms: conditions — HIV Infections | interventions — Enfuvirtide

INTERVENTIONS:
Drug: Enfuvirtide

SUMMARY:
The purpose of this study is to show if a dose of T-20 added to an anti-HIV combination (chosen specifically for each patient) lowers viral load by at least a certain level after 24 weeks as compared to an anti-HIV combination (chosen specifically for each patient) alone. Another purpose is to show if the patient response to T-20 will be maintained for 48 weeks.

DETAILED DESCRIPTION:
An OB regimen is selected to be initiated at baseline by the physician and patient. The OB regimen is based on the patient's prior treatment history as well as the results from the first screening visit HIV-1 genotypic and phenotypic (GT and PT) resistance testing and prior GT/PT antiretroviral resistance testing (if available). Prior or current laboratory abnormalities, including triglycerides and cholesterol, should also be taken into account when selecting the OB regimen. Patients are stratified with respect to the following: 1) screening viral load (less than 40,000 or 40,000 or more copies/ml); and 2) number of allowed investigational antiretrovirals (0, 1, or 2). Patients then are randomized to receive 1 of the following treatments for 48 weeks: OB regimen or OB plus T-20 regimen. Patients are seen for evaluation of efficacy and safety at Weeks 1, 2, and 4, every 4 weeks through Week 24, and then every 8 weeks through Week 48. In addition, efficacy only is evaluated at Weeks 6, 10, and 14. Patients also may be seen at additional visits during the study for plasma HIV-1 RNA measurements to potentially confirm virological failure.

Patients initially randomized to the OB arm who meet the criteria for virological failure and who switch to OB plus T-20 after Week 8 are followed under a new ("switch") schedule of assessments. Patients are encouraged to change their OB regimen at the time of switch.

Patients initially randomized to the OB plus T-20 arm who meet the criteria for virological failure may continue to receive OB plus T-20 if the patient and the physician feel that there is sufficient benefit. Patients are encouraged to change their OB regimen after Week 8 if they choose to continue on OB plus T-20 despite meeting the criteria for virological failure.

Patients on OB or OB plus T-20 arm who meet the criteria for virological failure but who do not wish to either switch to T-20 (for patients initially randomized to OB arm) or continue with T-20 (for patients initially randomized to OB plus T-20) are allowed to remain in the study for a maximum of 1 month.

At the end of the 48 weeks of treatment, patients are allowed to participate in 1 of the following treatment extensions: a) roll-over and receive OB plus T-20 (for patients receiving OB alone); or b) continue taking OB plus T-20 (for patients already receiving OB plus T-20), for a maximum of an additional 48 weeks (plus 4 weeks safety follow-up period), or until 12 weeks after commercial availability of T-20 in the country in which they are treated, whichever comes first. All patients are followed for a maximum of 100 weeks from their initial baseline visit date.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV infected.
* Are at least 16 years of age.
* Have an HIV-1 RNA of at least 5,000 copies/ml.
* Have received anti-HIV drugs for at least 3 months and/or have written records of resistance to at least 1 member of each of the 3 classes of anti-HIV drugs (nucleoside reverse transcriptase inhibitors [NRTIs], nonnucleoside reverse transcriptase inhibitors [NNRTIs], and protease inhibitors [PIs]). Resistance to NNRTIs may not be required in certain cases.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 525

CONTACTS AND LOCATIONS:
Locations (37):
- Australia (7):
  - Carlton Clinic, Carlton
  - Holdsworth House General Practice, Darlinghurst
  - Saint Vincent's Hosp, Darlinghurst
  - Royal Brisbane Hosp, Herston
  - Alfred Hosp, Prahan
  - Prahran Market Clinic, South Yarra
  - Taylors Square Clinic, Sydney
- Belgium (3):
  - Inst of Tropical Medicine, Antwerp
  - CHU Saint Pierre, Brussels
  - UZ Gasthuisberg, Leuven
- Germany (4):
  - Rheinische Friedrich Wilhelms Universitaet Medizinische, Bonn
  - Klinikum Der Johann Wolfgang Goethe Universitat, Frankfurt
  - Allgemeines Krankenhaus St Georg, Hamburg
  - Universitatskrankenhaus Eppendorf, Hamburg
- Italy (3):
  - UO Malattie Infettive, Florence
  - Clinica Malattie Infettive, Milan
  - Ospedale Amedeo di Savoia, Torino
- Netherlands (2):
  - Natac Med Centre, Amsterdam
  - Univ Medical Center Utrecht, CX Utrecht
- Spain (3):
  - Hospital Germans Trias I Pujol, Barcelona
  - Hosp La Paz, Madrid
  - Hospital General Universitario, Valencia
- Sweden (3):
  - University Hospital Mas, Malmo
  - Karolinska Hospital, Stockholm
  - Venhalsan Soder Hosp, Stockholm
- Switzerland (4):
  - Univ Hosp Basel / Med Outpatient Dept, Basel
  - Hopital cantonal / Div des maladies infectieuses, Geneva
  - CHUV, Lausanne
  - Universitatsspital Zurich, Zurich
- United Kingdom (8):
  - Brighton Gen Hosp, Brighton
  - Western Gen Hosp, Edinburgh
  - Royal Liverpool Univ Hosp, Liverpool
  - Chelsea and Westminster Hosp, London
  - King's College Hospital, London
  - Royal Free Hosp, London
  - Univ College London Med School, London
  - North Manchester Gen Hosp, Manchester

REFERENCES:
- [Background] Lazzarin A, Clotet B, Cooper D, Reynes J, Arasteh K, Nelson M, Katlama C, Stellbrink HJ, Delfraissy JF, Lange J, Huson L, DeMasi R, Wat C, Delehanty J, Drobnes C, Salgo M; TORO 2 Study Group. Efficacy of enfuvirtide in patients infected with drug-resistant HIV-1 in Europe and Australia. N Engl J Med. 2003 May 29;348(22):2186-95. doi: 10.1056/NEJMoa035211. PMID 12773645